CLINICAL TRIAL: NCT05337995
Title: Locomotion Strategies of Patients With Chronic Non-Specific Low Back Pain During Aperture Crossing
Brief Title: Locomotion Strategies of Low Back Pain Patients
Status: Completed | Type: Observational
Sponsor: University of Rennes 2 (Other)
Responsible Party: Principal Investigator, Agathe Bilhaut, PhD Student, University of Rennes 2
Other Study IDs: PERL
Record Dates: First submitted 2022-03-30; First posted 2022-04-20 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Chronic Low-back Pain; Walking
Keywords: Low Back Pain; Psychomotor Performance / physiology; Walking / physiology*; Adult; Humans; Motion Perception / physiology*
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Specific Low Back Pain patients: Participants must have pain located between the thoracolumbar hinge and the lower gluteal fold, with or without pain in either leg, present for more than 12 weeks, on a daily or almost daily basis (at least 4 days out of 7).
  Interventions: Other: Quantified analysis of walking during a task of passage through a horizontal opening
- Control group: Participant with no current or past chronic pain
  Interventions: Other: Quantified analysis of walking during a task of passage through a horizontal opening

INTERVENTIONS:
Other: Quantified analysis of walking during a task of passage through a horizontal opening — Functional test that reproduce a task of daily living, similar to a doorway

SUMMARY:
The biomechanical parameters studied in non-specific chronic low back pain patients in a locomotion task have so far focused on straight line walking. Although locomotion is primarily an automated action composed of repetitive patterns allowing movement from one place to another, walkers must respond to the environmental demands.These modifications show a flexible and adaptive approach to the constraints of the environment. In this study, we are particularly interested in a task of passage through a horizontal opening, similar to a doorway, which is a standardized task that has shown its interest in the study of perceptual-motor co-ordinations. In particular, it allows to consider anthropometric and functional abilities of individuals, reflecting their action capacities.

ELIGIBILITY:
Inclusion Criteria NSCLBP patients:

* Participants must have pain located between the thoracolumbar hinge and the lower gluteal fold, with or without pain in either leg.
* This pain must have been present for more than 12 weeks, on a daily or almost daily basis (at least 4 days out of 7)
* Participants must not be on any treatment or have been on stable analgesic treatment for at least 2 weeks prior to inclusion
* Participants must speak, read and understand French
* Participants must be between 18 and 65 years of age
* Participants must be able to understand simple commands and experimental instructions
* Participants must have normal or corrected vision
* Participants must have given informed consent to participate in the study
* Participants must be enrolled in or receiving social security benefits

Exclusion Criteria NSCLBP patients:

* Participants must not be pregnant or nursing mothers.
* Participants must not have cognitive or psychological impairments that are incompatible with compliance and/or understanding of the protocol (MMSE > 28)
* Participants must not be unable to understand informed consent, or be under guardianship or conservatorship
* Subjects must not already be participating in another research protocol involving the human subject or in parallel
* Participants must not be persons deprived of liberty by judicial or administrative decision
* Participants must not be under psychiatric care
* The participants must not present neurological signs evoking a neurodegenerative disease responsible for walking disorders (parkinsonian syndrome, ...)
* The participants must not present warning signs (red flags) pointing to an underlying pathology requiring specific and/or urgent care such as

  1. Ongoing litigation following a work-related accident
  2. Pain related to a cancer diagnosis
  3. Associated spinal cord symptoms (pyramidal signs, coordination disorders, motor or sensory deficits, sphincter disorders, etc.)
  4. Pain following an infection (night sweats, fever, chills, intravenous drug abuse, immunodeficiency, recent surgery, urinary or skin infection, etc.)
  5. Recent or pathological fractures (traffic accidents, history of osteoporosis, chronic use of corticosteroids, advanced age, unexplained weight loss, fatigue, history of cancer, etc. )
  6. Vascular problems (cold feet, decreased peripheral arterial pulse, etc.)

Inclusion and Exclusion Criteria of control group :

Participants strictly meet the same inclusion and non-inclusion criteria as NSCLBP patients, but must not have ongoing chronic pain or a history of significant chronic pain (≥ 4/10 for at least 6 months). They are matched for age and gender. They must not have any pathologies that affect walking or posture. These individuals must be able to perform the studied movements without the appearance of discomfort or exaggerated fatigue.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NSCLBP patients who do their medical follow-up in medical center in France
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Critical threshold | Clinical assessment at base line
  Defined as the width of opening making the transition between openings that it is possible or not to cross while walking without modification of the movement. We will then identify the trials, i.e. the door widths, where the participants have turned their shoulders. To do this, we will compare the shoulder angle observed during the doorway crossing with the average angle observed in the control conditions, corresponding to a straight line walk without any opening to cross.

SECONDARY OUTCOMES:
Phase shift between shoulder and pelvic angles in the transverse plane | Clinical assessment at base line
  Analysis of the difference between the scapular and pelvic angles in the transverse plane during aperture crossing
Stability of the trunk | Clinical assessment at base line
  Analysis of the amplitude of the medio-lateral oscillation movements in the frontal plane during the task
Step length | Clinical assessment at base line
  Analysis of the step length before the obstacle compared to the step length in the nominal walking condition (with no obstacle in the path)
Walking speed | Clinical assessment at base line
  Analysis of the walking speed before the obstacle compared to the walking speed in the nominal walking condition (without obstacle on the path)

OTHER OUTCOMES:
Pain intensity | Clinical assessment at base line
  Pain intensity reflects the overall magnitude of the patient's perceived pain experience. We will assess this variable using a visual analogue scale (VAS) in paper format. The VAS is represented by a 100 mm long horizontal line with descriptors at both ends: on the left "no pain" and on the right "worst pain imaginable". The patient must then draw a mark on the line corresponding to his or her pain experience. "0" corresponds to "no pain" and "10" corresponds to "worst pain imaginable".
Temporal aspects of pain | Clinical assessment at base line
  Assessment of the impact of the variability of pain over time, i.e. the duration of painful episodes (in number of months).
Levels of anxiety and depression | Clinical assessment at base line
  Anxiety refers to fear, extreme worrying and hyperarousal symptoms. Depression refers to negative mood, loss of self-confidence, loss of motivation and pleasure. We will use these measures using the Hospital Anxiety Depression Scale (HADS). This tool consists of 14 items scored from 0 to 3. Seven questions relate to anxiety (Total A) and 7 questions to the depressive dimension (Total D), resulting in two scores with a maximum total of 21 each. The higher the score, the more anxiety or depression the person has.
Pain Catastrophizing | Clinical assessment at base line
  Catastrophizing refers to the cognitive process in which anxious patients dwell on the most negative consequences and refers here to the interpretation of pain as extremely threatening. We will use the Pain Catastrophizing Scale (PCS) to assess three dimensions: rumination, amplification and helplessness. This scale consists of 13 items scored from 0 (not at all) to 4 (all the time) with a maximum score of 52. The higher the score, the greater the level of catastrophisation.
Kinesiophobia | Clinical assessment at base line
  Fear of movement is characterized by pain-related fears and anxieties that often result in avoidance of movement that could cause or worsen an injury. We will use the Tampa Scale Kinesiophobia (TSK). This scale consists of 17 items rated from 1 (strongly disagree) to 4 (strongly agree) with a maximum score of 68. The higher the score, the greater the level of kinesiophobia.
Psychological Inflexibility in Pain | Clinical assessment at base line
  Psychological flexibility measures psychological functioning in phase (in fusion) with the pain or whether the patient has certain degrees of freedom from it. We will use the Psychological Inflexibility in Pain Scale (PIPS) allowing us to assess two factors: avoidance and cognitive fusion. This scale consists of 16 items with a scale of 1 (never true) to 7 (always true). The higher the score, the greater the level of psychological inflexibility.
Fear Avoidance Beliefs | Clinical assessment at base line
  Fear and avoidance beliefs reflect patients' pain avoidance behaviors. We will use the Fear Avoidance Beliefs Questionnaire (FABQ) to assess two subscales: beliefs about work and beliefs about physical activity. The questionnaire consists of 16 items scored from 0 (absolutely disagree with the sentence) to 6 (completely agree with the sentence). The maximum score for beliefs about work is 42 and the maximum score for beliefs about physical activity is 24. The higher the score, the greater the level of beliefs.
Physical functioning | Clinical assessment at base line
  Physical functioning refers to the impact on the patient's ability to perform daily physical activities necessary to meet basic needs, ranging from self-care to more complex activities that require a combination of skills. We will use the Roland Morris Disability Questionnaire (RMDQ). This questionnaire has 24 items with a maximum score of 24. The higher the score, the more functional disabilities the person has.
Quality of life (EQ-5D) | Clinical assessment at base line
  Quality of life refers to the impact on the physical, psychological, and social domains of health, considered as distinct domains that are influenced by a person's experiences, beliefs, expectations, and perceptions. We will use the EuroQol 5 Dimension questionnaire (EQ-5D) allowing for the assessment of five dimensions: mobility, ability to care for oneself, usual work, home, and leisure activities, pain/discomfort, anxiety, and depression. Five degrees of severity in ascending order are used to assess each dimension: "no problems" to "total disability" for items that assess ability, and "no problem" to "extreme" for the other items. The higher the score, the lower the level of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Roze, MD, Principal Investigator — clinique de la Sagesse
Locations (1):
- University of Rennes 2, Rennes, France

REFERENCES:
- [Derived] Bilhaut A, Menard M, Roze O, Cretual A, Olivier AH. Locomotion behavior of chronic Non-Specific Low Back Pain (cNSLBP) participants while walking through apertures. Gait Posture. 2023 Jul;104:140-146. doi: 10.1016/j.gaitpost.2023.06.015. Epub 2023 Jun 22. PMID 37419055